CLINICAL TRIAL: NCT03046654
Title: Cervical Cerclage Position Throughout Pregnancy, it's Distance From the Inner and Outer Cervical os', and Implications of the Position on Pregnancy Outcomes.
Brief Title: Cervical Cerclage Position Throughout the Pregnancy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in patient recruitment
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0247-15-RMB
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cervix Uteri-Diseases
MeSH Terms: interventions — Gynecological Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical cerclage (Experimental): Women with a poor obstetric history that require cervical cerclage in order to avoid late abortion/early delivery.
  Interventions: Diagnostic Test: Trans vaginal sonography; Diagnostic Test: Vaginal examination; Diagnostic Test: Speculum examination

INTERVENTIONS:
Diagnostic Test: Trans vaginal sonography — Trans vaginal sonography performed once every 4 weeks from the time of cerclage placement until the time of cerclage removal to evaluate cerclage position and distance from internal and external os'.
Diagnostic Test: Vaginal examination — Vaginal examination performed once every 4 weeks from the time of cerclage placement until the time of cerclage removal to evaluate cervical conditions including cervical dilatation, cervical effacement and pressure on the cerclage.
Diagnostic Test: Speculum examination — Speculum examination performed once every 4 weeks from the time of cerclage placement until the time of cerclage removal to evaluate cerclage position and vaginal bleeding.

SUMMARY:
Cervical cerclage is an obstetric intervention used in women with poor obstetric histories. After recruiting the participant, Trans vaginal sonography will be used to examine cervical length and funneling. In addition vaginal examination will be performed to evaluate the cervix. After placing the cerclage, the participant will be invited every 4 weeks for a follow up evaluation session in order to examine the cervix and cerclage position. .

DETAILED DESCRIPTION:
Cervical cerclage is an obstetric intervention used in women with poor obstetric histories due to late abortions, premature deliveries and painless dilatation. These 3 situations are usually due to cervical incompetence though can be caused by infection and other factors.

The cerclage is usually placed from 12-24 weeks of gestation depending on the indication and medical follow up during pregnancy. There are 2 methods for cerclage performance-McDonald and Shirodkar that have the same efficacy.

After recruiting the participant, Trans vaginal sonography will be used to examine cervical length and funneling. In addition vaginal examination will be performed to evaluate the cervix. After placing the cerclage, the participant will be invited every 4 weeks for a follow up evaluation session in order to examine the cervix and cerclage position. Each follow up will include a vaginal examination and trans vaginal sonography. The trans vaginal sonography will examine total cervical length, funneling, and the cerclage's distance from the inner and outer os' of the cervix.

ELIGIBILITY:
Inclusion Criteria:

* Women that have a cervical cerclage placed during pregnancy at the investigator's medical center.

Exclusion Criteria:

* Women that do not require cervical cerclage.
* Women that had a cervical cerclage placed at a different medical center.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 7 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Gestational age at the time of delivery | Up to 9 months
  Gestational age at the time of delivery

SECONDARY OUTCOMES:
Gestational age at the time of the removal of the cervical cerclage | Up to 9 months
  Gestational age at the time of the removal of the cervical cerclage

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No